CLINICAL TRIAL: NCT06169046
Title: A Placebo-controlled Study to Evaluate the Efficacy and Safety of Clenbuterol in Patients With Spinal and Bulbar Muscular Atrophy (SBMA)
Brief Title: A Placebo-controlled Study of Clenbuterol in Spinal and Bulbar Muscular Atrophy
Acronym: BetaSBMA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gianni Soraru (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor-Investigator, Gianni Soraru, Professor, University Hospital Padova
Organization: University Hospital Padova (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT: 2017-005103-27
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Spinal and Bulbar Muscular Atrophy
Keywords: SBMA; clenbuterol; trial
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked | interventions — Clenbuterol; Exercise

STUDY DESIGN:
Intervention Model Description: 2 parallel groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clenbuterole (Experimental): 45 patients will receive Clenbuterol at a final dosage of 0.04 mg/day, treated for a total of 48 weeks
  Interventions: Drug: Clenbuterol
- placebo (Placebo Comparator): 45 patients will receive placebo, treated for a total of 48 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clenbuterol — tablets
  Other Names: active
  Arms: clenbuterole
Drug: Placebo — tablets
  Arms: placebo

SUMMARY:
There is no cure to arrest or delay SBMA progression. It is estimated that ~1000 individuals are affected by SBMA in Italy at any given time (prevalence: 1.5/100000) with an annual incidence of 0.19/100000 males. Here, we are going to test the potential of beta2-agonist stimulation on muscle as a therapeutic avenue for SBMA. We have provided pre-clinical evidence that β-agonist stimulation may be a therapeutic strategy for SBMA. Moreover, we have shown that beta2-agonists are effective in improving motor function without relevant adverse events in a small cohort of SBMA patients. To establish safety and efficacy of clenbuterol as a cure for SBMA, we are conducting a multicenter, phase II, randomized, double-blind, parallel-group, single dose, placebo-controlled trial. Indeed, based on our preliminary data, some concerns remain to be addressed.

ELIGIBILITY:
Inclusion Criteria:

1. males who have received a genetically confirmed diagnosis of SBMA (AR CAG repeat number >= 38);
2. aged between 18 and 75 (+364 days) years;
3. displaying one or more of the following clinical symptoms: muscle atrophy, limb weakness, bulbar palsy;
4. able to walk independently with or without a cane or other supporting device (all supporting devices are acceptable except on wheelchair);
5. providing a written informed consent.

Exclusion Criteria:

1. a documented cardiovascular disease precluding the use of beta2 agonists (in the judgment of the investigators);
2. glaucoma, severe prostatic hypertrophy, hyperthyroidism, pheochromocytoma, and other medical conditions that, in the judgment of the investigators, would expose the patient to undue risk of harm or prevent the patient from completing the study;
3. concomitant treatment with either beta-blockers or sympathomimetic drugs (If a beta-blockers concomitant medication is ongoing before the study inclusion, the patient can be enrolled if the beta-blocker is discontinued for 3 weeks prior to randomization visit);
4. inability to walk or walking only with the support of a caregiver;
5. use of beta2 agonists in the preceding 6 months;
6. participation to an interventional trial in the preceding 3 months;
7. neuromuscular disease other than SBMA.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
6-minute-walk test | 48 weeks
  to assess the efficacy of chronic treatment with clenbuterol in patients with SBMA by the 6MW test

SECONDARY OUTCOMES:
SBMA-FRS scale | 48 weeks
  SBMA-FRS total score during the 12-months treatment period (from V2 to V7) in the two treatment arms
Adult Myopathy Assessment Tool (AMAT) | 48 weeks
  AMAT total score during the 12-months treatment period (from V2 to V7) in the two treatment arms
FVC | 48 weeks
  FVC during the 12-months treatment period (from V2 to V7) in the two treatment arms
6K scale | 48 weeks
  6K total score during the 12-months treatment period (from V2 to V7) in the two treatment arms
Serum creatinine levels | 48 weeks
  serum creatinine levels during the 12-months treatment period (from V2 to V7) in the two treatment arms
ALSAQ-40 | 48 weeks
  ALSAQ-40 total score during the 12-months treatment period (from V2 to V7) in the two treatment arms
individualized neuromuscular quality of life (INQoL) questionnaire | 48 weeks
  INQOL total score during the 12-months treatment period (from V2 to V7) in the two treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Gianni Sorarù, MD, Principal Investigator — Azienda Ospedale Università di Padova
Locations (1):
- Azienda Ospedale Università di Padova, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: Undecided